CLINICAL TRIAL: NCT06416410
Title: An Open-label, Randomized, Positive Control, Multicenter Phase III Clinical Study. Evaluating JAB-21822 Combined With JAB-3312 Compared Tislelizumab Combined With Pemetrexed + Carboplatin in the First Line for Treatment of Advanced Non-squamous Non-small Cell Lung Cancer With KRAS p.G12C Mutation
Brief Title: JAB-21822 Combined With JAB-3312 Compared SOC in the First Line for Treatment of Advanced Non-small Cell Lung Cancer With KRAS p.G12C Mutation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-3002
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer; Metastatic Non-squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — tislelizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JAB-21822+JAB-3312 (Experimental): JAB-21822 tablet, 21 days as a treatment cycle; JAB-3312 tablet/capsule, 21 days as a treatment cycle
  Interventions: Drug: JAB-21822; Drug: JAB-3312
- Tislelizumab combined with Pemetrexed + Carboplatin (Active Comparator): Tislelizumab injection, 21 days as a treatment cycle; Pemetrexed injection, 21 days as a treatment cycle; Carboplatin injection, 21 days as a treatment cycle
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: JAB-21822 — JAB-21822 administered orally as a tablet
  Arms: JAB-21822+JAB-3312
Drug: Tislelizumab — Tislelizumab administered as an intravenous (IV) infusion
  Arms: Tislelizumab combined with Pemetrexed + Carboplatin
Drug: JAB-3312 — JAB-3312 administered orally as a tablet or capsule
  Arms: JAB-21822+JAB-3312
Drug: Pemetrexed — Pemetrexed administered as an intravenous (IV) infusion
  Arms: Tislelizumab combined with Pemetrexed + Carboplatin
Drug: Carboplatin — Carboplatin administered as an intravenous (IV) infusion
  Arms: Tislelizumab combined with Pemetrexed + Carboplatin

SUMMARY:
This Phase 3 study will evaluate the efficacy of JAB-21822+JAB-3312 versus tislelizumab (PD-1 Ab) combined with pemetrexed+carboplatin as the first line treatment in subjects with KRAS G12C mutated locally advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* A signed written informed consent is required before performing any study-related operations
* Age greater than or equal to 18 years old
* Histologically or cytologically confirmed locally advanced/metastatic, unresectable non-squamous NSCLC with KRAS p. G12C mutation confirmed by the central lab
* No history of systemic anticancer therapy to the local advanced/metastatic disease
* Expected survival period greater than or equal to 3 months
* Having at least one target lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) ≤ 1

Exclusion Criteria:

* Previous (≤2 years) or current solid tumors or hematologic tumors of other pathological types
* Carry other driver gene mutations with available target therapy, or carry other KRAS mutations
* Subjects with untreated central nervous system (CNS) metastases were excluded;
* Uncontrolled pleural effusion, pericardial effusion, and ascites
* Subjects with impaired heart function or clinically significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Outcome Progression-free Survival (PFS) | From Baseline up to 4 years
  PFS is defined as the time from randomization until the first documentation of radiologic disease progression or death due to any cause, whichever occurs first. Progression will be based on Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, per Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From Baseline up to 4 years
  Objective response is defined as the best overall response of complete response (CR) or partial response (PR), based on RECIST v1.1
Overall Survival (OS) | From Baseline up to 4 years
  OS is defined as the time from randomization until death due to any cause
Number of Participants With Treatment-Emergent Adverse Events | From Baseline up to 4 years
Number of Participants With Clinically Significant Changes in Vital Signs | From Baseline up to 4 years
Time to Maximum Plasma Concentration (Tmax) | Pre-dose Day 1 up to Day 64
Half life (t1/2) | Pre-dose Day 1 up to Day 64

OTHER OUTCOMES:
Patient Self-Evaluation Results (PRO) | From Baseline up to 4 years
  To be assessed by EORTC OLO-LC13
Patient Self-Evaluation Results (PRO) | From Baseline up to 4 years
  To be assessed by EORTC OLO-C30
Patient Self-Evaluation Results (PRO) | From Baseline up to 4 years
  To be assessed by EuroQoL(EQ)5D

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jie M.D., Principal Investigator — Cancer Institute and Hospital
Locations (37):
- China (37):
  - Anhui Province cancer hospital, Hefei, Anhui
  - Pecking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy Of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Captal Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Fujian cancer Hospital, Fuzhou, Fujian
  - The first Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy Of medical Sciences Shenzhen Center, Shenzhen, Guangdong
  - Guangxi Medical University Cancer hospital & Guangxi Cancer Institute, Nanning, Guangxi
  - Cangzhou hospital of integrated TCM-WM Hebei, Cangzhou, Hebei
  - Harbin Medical University Cancer Hospital-Mammary gland of internal, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hosipital Of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Hubei cancer hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jilin cancer hospital, Jilin, Jilin
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - The affiliated hospital of Qingdao university, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi province cancer hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - Sichuan province cancer hospital, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute Hospital, Tianjin, Tianjin Municipality
  - The First affiliated hospital Zhejiang university school of medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No